CLINICAL TRIAL: NCT00292799
Title: A Randomised Controlled Clinical Trial of Metformin Versus Orlistat for the Management of Obese Anovulatory Women.
Brief Title: An RCT of Metformin Vs Orlistat in Obese Anovulatory Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH14007
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Anovulation; Obesity
Keywords: Polycystic ovary syndrome; Obesity; metformin; orlistat
MeSH Terms: conditions — Anovulation; Obesity; Polycystic Ovary Syndrome

INTERVENTIONS:
Drug: Orlistat Vs Metformin

SUMMARY:
This study aims to investigate the role of the weight reduction agent, Orlistat compared to the Metformin for the management of women who are obese and do not ovulate or have difficulty conceiving. Patients will receive either one of these medications and will be monitored at regular intervals with hormone blood tests and ultrasound scans in order to study the effect of the medications on the reproductive functions. Patients will receive the medications for three months and the study will end if the patient becomes pregnant. The study also aims to investigate the dose of metformin that should be used as there is no consensus to date regarding the optimum dosage for this drug

DETAILED DESCRIPTION:
We aim to recruit 40 patients suffering from anovulatory obesity with a BMI of 30 or more. Patients will be included from all ethnic groups.

Patients will have a baseline history, clinical examination, hormonal profile (FSH/LH, fasting Insulin/glucose ratio, androgen profile, day 21 serum progesterone, serum leptin and ghrelin levels) ultrasound examination (ovarian volume and antral follicle count), including Doppler blood flow study (ovarian stromal velocity, PI, RI, SD ratio and power Doppler) Participants will then be randomised to receive either metformin or orlistat. Patients receiving orlistat will receive the standard dose of the drug as recommended in the BNF. Metformin will be given in an incremental dose starting at 1000mg per day and increased at 4 weekly intervals to 2000mg/d, depending on the occurrence of any gastrointestinal intolerance. The endocrinological and ultrasound investigations will be repeated at 4 weekly intervals. Both groups will be given a standard exercise and diet program in conjunction with medical treatment.

The clinical endpoint will be the achievement of conception, a Body Mass Index of less than 30, or completion of a 3-month course of treatment.

Study design:

A randomised controlled open label clinical trial. Participants be randomised using a computer generated randomisation program available at the pharmacy of the Jessop Wing, into either one of two arms: metformin or orlistat. The randomisation will be stratified in order to achieve a homogenous distribution of PCOS and non-PCOS patients in both arms of the study.

ELIGIBILITY:
Inclusion Criteria:

1. In the childbearing period 2. Obese with a body mass index of 30 or more. 3. Are anovulatory as shown by day 21-serum progesterone. 4. Polycystic ovarian syndrome will be diagnosed according if at least two of the following three features are present, after exclusion of other aetiologies (Azziz, 2004): (i) Oligo- or anovulation, (ii) Clinical and/or biochemical hyperandrogenism (iii) Polycystic ovaries.

Exclusion Criteria:

1. BMI of less than 30
2. Patients not requesting treatment for their symptoms
3. Patients with contraindications for any of the medications: renal or hepatic impairment, malabsorption syndrome, cholestasis
4. Diabetic patients
5. Pregnancy
6. Breast feeding

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Outcome measures:
1- The occurrence of ovulation as measured by day-21 serum progesterone ( equal to or more than 30mmol/L).
2- Number of patients who have lost at least 5% of body weight at the end of the study.
3- Improvement/deterioration of clinical symptoms: hyper androgenic features, obesity and menstrual disturbances
4- Change in the ovarian Doppler indices.

CONTACTS AND LOCATIONS:
Overall Officials: Professor William L Ledger, D.Phil,FRCOG, Study Chair — Sheffield University; Dr Mostafa Metwally, Study Director — Sheffield University; Professor TC Li, Study Chair — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Trust, Jessop Wing, Sheffield, United Kingdom

REFERENCES:
- [Derived] Metwally M, Amer S, Li TC, Ledger WL. An RCT of metformin versus orlistat for the management of obese anovulatory women. Hum Reprod. 2009 Apr;24(4):966-75. doi: 10.1093/humrep/den454. Epub 2008 Dec 18. PMID 19095663